CLINICAL TRIAL: NCT03447613
Title: Association of Retinal Nerve Fiber Layer (RNFL) Thickness With Cerebrospinal Fluid Aβ and Tau Concentration
Brief Title: Retinal Nerve Fiber Layer Thickness and Cerebrospinal Fluid Aβ/Tau
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yuan Shen, MD, PhD, Chief of Psychiatry Department, Shanghai 10th People's Hospital
Other Study IDs: dsyy001
Record Dates: First submitted 2018-02-17; First posted 2018-02-27 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Alzheimer Disease
Keywords: retinal nerve fiber layer; cerebrospinal fluid Aβ and Tau
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1 ml of CSF was collected from a spinal needle by anesthesiologists during the spinal anesthesia before the administration of the local anesthetic. The CSF was collected in an Eppendorf tube and was immediately stored in a -80 °C degree freezer until the time of measurement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly participants with surgery: The studied cohort were participants 50 years old or older, without a diagnosis of dementia, and scheduled to have orthopedic or urological surgery under spinal anesthesia at Shanghai 10th People's Hospital.
  Interventions: Procedure: surgery

INTERVENTIONS:
Procedure: surgery — All participants were scheduled to have elective total hip or knee replacement surgery, ureteroscopic lithotripsy and transurethral resection of the prostate under spinal anesthesia at the Shanghai 10th People's Hospital. After 5 years, the investigaors will follow up the participants including cognitive functions, PET-CT, thickness of Retinal Nerve Fiber Layer.

SUMMARY:
To test the hypothesis that retinal nerve fiber layer (RNFL) thickness is correlated with Aβ and Tau concentration of cerebrospinal fluid (CSF) in an older population.

DETAILED DESCRIPTION:
retinal nerve fiber layer (RNFL) thickness changing has been reported in Alzheimer's Disease (AD) patients at an early stage, and has been demonstrated as a potential biomarker able to predict cognitive deterioration (Hinton DR et al., N Engl J Med 1986; London A et al. Nat Rev Neurol 2013; Chang LY et al., Alzheimers Dement 2014). However, whether RNFL thickness is correlated with cerebrospinal fluid (CSF) features of AD pathogenesis (e.g., Aβ and Tau) remains unclear. The investigators thus conducted this observational cohort study to test the correlation between RNFL thickness changing and CSF, to further validate RNFL as a potential AD biomarker.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years old or older;
2. five years or more of education and scores of MMSE ≥ 24 points;
3. Chinese as their first language;
4. Having spinal anesthesia.

Exclusion Criteria:

1. prior diagnoses of neurologic diseases, e.g., dementia, Parkinson's diseases, multiple sclerosis or stroke according to DSM-IV;
2. history of mental disorders (e.g., major depressive disorder and schizophrenia) diagnosed according to DSM-IV;
3. known diseases contributing to the retina pathologies, e.g., diabetes, glaucoma or increased intraocular pressure (more than 22 mmHg), cataract, and macular degeneration and hypermyopia;
4. unwillingness to comply with the cognitive assessments;
5. ungradable images of OCT.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 300 old adults who were scheduled to have elective total hip or knee replacement surgery, ureteroscopic lithotripsy and transurethral resection of the prostate at the Shanghai 10th People's Hospital were asked to participate in this study. A total of 104 participants were enrolled from August 2013 to December 2014, and the data from 86 participants were finally included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Specific cognitive function | Within one week before surgery
  Neuropsychological test battery to assess specific cognitive function, including immediate memory, visuospatial memory and executive function.

SECONDARY OUTCOMES:
retinal nerve fiber layer (RNFL) thickness | Within one week before surgery
  Optical coherence tomography (Carl Zeiss Meditec, Inc., Dublin, CA, USA) to measure RNFL thickness
Cerebrospinal fluid (CSF) Aβ concentration | During the spinal anesthesia before the administration of the local anesthetic.
  ELISA kits (Aβ40: Cat. # 292-62301; Aβ42: Cat. # 296-64401, Wako, Richmond, VA) to measure Aβ concentration
Cerebrospinal fluid (CSF) Tau concentration | During the spinal anesthesia before the administration of the local anesthetic.
  ELISA kits (Tau: Cat. # KHB0041, Invitrogen, San Francisco, CA) to measure Aβ concentration
Global cognitive state | Within one week before surgery
  Mini-Mental State Examination (MMSE) to assess global cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Shen, MD, PhD, Principal Investigator — Shanghai 10th People's Hospital
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] London A, Benhar I, Schwartz M. The retina as a window to the brain-from eye research to CNS disorders. Nat Rev Neurol. 2013 Jan;9(1):44-53. doi: 10.1038/nrneurol.2012.227. Epub 2012 Nov 20. PMID 23165340
- [Result] Chang LY, Lowe J, Ardiles A, Lim J, Grey AC, Robertson K, Danesh-Meyer H, Palacios AG, Acosta ML. Alzheimer's disease in the human eye. Clinical tests that identify ocular and visual information processing deficit as biomarkers. Alzheimers Dement. 2014 Mar;10(2):251-61. doi: 10.1016/j.jalz.2013.06.004. Epub 2013 Sep 5. PMID 24011928
- [Result] Hinton DR, Sadun AA, Blanks JC, Miller CA. Optic-nerve degeneration in Alzheimer's disease. N Engl J Med. 1986 Aug 21;315(8):485-7. doi: 10.1056/NEJM198608213150804. PMID 3736630